CLINICAL TRIAL: NCT06777550
Title: The Feasibility of Using Simucase TM As Part of an Alternative Clinical Learning Method for Malaysian Health Sciences Education
Brief Title: Use of Simucase for Clinical Learning in Malaysia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Collaborators: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Farahiyah Wan Yunus, Principle Investigator and Head of Site Investigator, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: JEP-2024-967
Record Dates: First submitted 2025-01-08; First posted 2025-01-16 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Clinical Learning
Keywords: clinical; simucase; health science; education; alternative learning; rehabilitation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SimucaseTM (Active Comparator): The experiment group - who will receive the clinical learning method using SimucaseTM
  Interventions: Other: SimucaseTM
- Conventional clinical learning (Active Comparator): The control group - which will accept conventional clinical learning methods such as problem-based learning case-study case studies
  Interventions: Other: Conventional Clinical Learning

INTERVENTIONS:
Other: SimucaseTM — experiment group - who will receive the clinical learning method using SimucaseTM
  Arms: SimucaseTM
Other: Conventional Clinical Learning — Problem-based learning case-study case studies
  Arms: Conventional clinical learning

SUMMARY:
The goal of this feasibility study is to the investigate the use of Simucase in the context of health science learning in Malaysia. This study can be a catalyst for technology-based clinical learning than just conventional methods to enrich the learning experience. This can influence the policy in promoting the effective use of existing commercial technologies in clinical learning for health science programs in Malaysia and can transform national higher education scenario in the future.

An experimental study with 24 participants from the rehabilitation disciplines of audiology, occupational therapy, physiotherapy, and speech therapy method using a pilot study techniques of clinical control studies. Participants will be assigned to either the experimental group who will receive the clinical learning method using SimucaseTM or (ii) the control group - which will accept conventional clinical learning methods such as problem-based learning case-study case studies. The topic of learning is the same for both groups.

The study hypothesis includes:

* There is a significant difference on clinical skills between SimucaseTM and conventional approach of learning among health science students.
* There is a significant difference on students' satisfaction learning between SimucaseTM and conventional approach of learning among health science students.

DETAILED DESCRIPTION:
INTRODUCTION

In line with the changing agenda of the international paradigm that promotes the use of technology in the learning of health studies to overcome problems related to placement, logistics, human resources for supervision, patient aversion and creating a safe and conducive learning environment to form good competencies before stepping into clinical field learning. World bodies such as the World Federation Occupational Therapists allow the replacement of 20% of clinical field training to alternative clinical learning such as the use of technology and tele-health.

This study can be a catalyst for technology-based clinical learning than just conventional methods to enrich the learning experience. This can influence the policy in promoting the effective use of existing commercial technologies in clinical learning for health science programs in Malaysia and can transform national higher education scenario in the future.

PROBLEM STATEMENT

Education research in allied health especially rehabilitation, is more marginalized than medicine or nursing. This retards the advancement of teaching and learning strategies to optimize allied health education. Adopting knowledge from other fields such as medicine and nursing may be less fitting with the allied health education's needs. Therefore, it is essential to tailor the available learning strategies carefully to optimize their learning benefits according to the discipline's needs.

The clinical placement was reported to have missed a substantial learning opportunity due to a lack of theoretical application and weak teaching skills among clinicians. Having clinical simulation to supplement clinical placement was beneficial to optimize the gain from clinical learning as it was constructed on a solid learning theory. Simulation has become more advanced with the current availability of technology in combination with gaming elements. The combination of virtual simulation and gaming element creates substantial learning opportunity based on Kolb's experiential learning model.

RESEARCH OBJECTIVES

Main Objective

• To investigate the applicability of SimucaseTM software for clinical learning among health science students.

Specific Objectives

* To investigate the efficacy of SimucaseTM compared to conventional approach for clinical skills.
* To compare students' satisfaction on learning using SimucaseTM over conventional approach in clinical learning among health science students.
* To explore the feasibility of SimucaseTM as an alternative learning method for clinical learning among health science students.

Study design

The experimental study method used pilot study techniques, clinical control studies is proposed. This method is a high-quality technique to ensure the effectiveness of an intervention is credible.

Study samples

Students will be selected from the disciplines of audiology, occupational therapy, physiotherapy, and speech therapy at an institution. It is expected that 24 students (12 per control and experiment group) for each discipline will be recruited. Only second- to fourth-year students will be recruited, as first-year students have not yet taken any specialized courses in the program, making them unprepared for clinical learning.

Procedure

Each discipline will conduct RCT research separately to reduce the bias of differences between fields of study. Here, each RCT research will divide the students into two groups using sample random sampling, namely (i) the experiment group - who will receive the clinical learning method using SimucaseTM; and (ii) the control group - which will accept conventional clinical learning methods such as problem-based learning case-study case studies. The topic of learning is the same for both groups. It is recommended to have a learning session of two sessions for each group within a week. After the end of the study, the study participants will be evaluated for their performance by answering some survey forms (i.e., SLSQ). Only one data collection time is done (i.e., post-test) only. For ethical purpose, the control group and the experiment group will be cross-over (e.g., swap) on the learning approach to experience both approaches but not evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Students from rehabilitation-related academic programmes such as occupational therapy, physiotherapy, speech therapy and audiology.
* Students from undergraduate second to fourth year of the academic programme.

Exclusion Criteria:

• International students Students who are not willing to participate in this program during the semester break.

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-19 (Estimated); Primary Completion 2025-12-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
The Clinical Learning Environment Comparison Survey (CLECS 2.0) | One (1) week of post-intervention
  The survey consists of 29 multiple items across various subscales, each representing different aspects of the clinical learning environment, such as communication, critical thinking, and technical skills. Students rate their experiences on a 4-point Likert scale, (4 =well-met, 3 =met, 2 = partially met, 1 = not met) with a not applicable (NA) option. The overall score for each subscale is calculated by averaging the responses for that particular domain, providing insight into specific areas of strength or weakness in the learning environment. The total score is a sum or average of all the subscale scores, offering a comprehensive assessment of the clinical learning environment as perceived by the students. A higher score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Farahiyah Wan Yunus, Doctor of Philosophy, Principal Investigator — National University of Malaysia; Muhammad H Romli, Doctor of Philosophy, Study Director — Universiti Putra Malaysia
Locations (1):
- National University of Malaysia, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] World Federation of Occupational Therapists. (2020). COVID-19 and WFOT minimum education standards statement, 2020. Available: https://www.wfot.org/news/2020/covid-19-and-wfot-minimum-education-standards-statement
- [Background] Waseh S, Dicker AP. Telemedicine Training in Undergraduate Medical Education: Mixed-Methods Review. JMIR Med Educ. 2019 Apr 8;5(1):e12515. doi: 10.2196/12515. PMID 30958269
- [Background] Thomas A, Burns R, Sanseau E, Auerbach M. Tips for Conducting Telesimulation-Based Medical Education. Cureus. 2021 Jan 4;13(1):e12479. doi: 10.7759/cureus.12479. PMID 33552792
- [Background] Romli MH, Wan Yunus F, Cheema MS, Abdul Hamid H, Mehat MZ, Md Hashim NF, Foong CC, Hong WH, Jaafar MH. A Meta-synthesis on Technology-Based Learning Among Healthcare Students in Southeast Asia. Med Sci Educ. 2022 May 7;32(3):657-677. doi: 10.1007/s40670-022-01564-3. eCollection 2022 Jun. PMID 35573465
- [Background] Romli MH, Foong CC, Hong WH, Subramaniam P, Wan Yunus F. Restructuring education activities for full online learning: findings from a qualitative study with Malaysian nursing students during Covid-19 pandemic. BMC Med Educ. 2022 Jul 11;22(1):535. doi: 10.1186/s12909-022-03587-1. PMID 35821126
- [Background] Rezaee M, Rassafiani M, Khankeh H, Hosseini MA. Experiences of occupational therapy students in the first fieldwork education: a qualitative study. Med J Islam Repub Iran. 2014 Oct 11;28:110. eCollection 2014. PMID 25664311
- [Background] Praveen, C., Herur, S., Vashisht, S., Venkatesh, V. K. & Senapati, S. (2022). A comparative study on the suitability of virtual labs for school chemistry experiments. Journal of Emerging Investigators, 5(1), 1-9.
- [Background] Nelson, J. (2017). Using conceptual depth criteria: addressing the challenge of reaching saturation in qualitative research. Qualitative Research, 17(5), 554-570. https://doi.org/10.1177/1468794116679873
- [Background] Mattila, A., Martin, R.M., DeIuliis, E.D. (2020). Simulated fieldwork: A virtual approach to clinical education. Education Sciences, 10, 272. https://doi.org/10.3390/educsci10100272
- [Background] Leighton, K. (2015). Development of the Clinical Learning Environment Comparison Survey. Clinical Simulation in Nursing, 11(1), 44-51. doi:10.1016/j.ecns.2014.11.002
- [Background] Ingwersen K, Lyons N, Hitch D. Perceptions of fieldwork in occupational therapy. Clin Teach. 2017 Feb;14(1):55-59. doi: 10.1111/tct.12518. Epub 2016 Apr 5. PMID 27060287
- [Background] Foronda CL, Fernandez-Burgos M, Nadeau C, Kelley CN, Henry MN. Virtual Simulation in Nursing Education: A Systematic Review Spanning 1996 to 2018. Simul Healthc. 2020 Feb;15(1):46-54. doi: 10.1097/SIH.0000000000000411. PMID 32028447
- [Background] Emslie B. Clinical occupational therapists' experience of their role as clinical educators during the fieldwork experience of occupational therapy students (master's thesis). South Africa, Stellenbosch University, Stellenbosch; (2012).
- [Background] DeIuliis, E., Mattila, A., & Martin, R. (2021). Level I FW in a simulated environment: A blueprint on how to use SimucaseTM. Journal of Occupational Therapy Education,5(2). Retrieved from https://encompass.eku.edu/jote/vol5/iss2/15/